CLINICAL TRIAL: NCT04921228
Title: Heart Rate Variability Biofeedback in Healthcare Providers During COVID-19: A Pilot Feasibility Study
Brief Title: Biofeedback for CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2021-233
Record Dates: First submitted 2021-05-20; First posted 2021-06-10 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Disordered Eating; Stress
Keywords: Heart rate variability biofeedback; Disordered eating; Eating Disorders; Perceived Stress; Interoception; Interoceptive awareness; Vagal tone; Mind-body approaches; Self-compassion; Resilience; Body appreciation; Self-care; Intuitive eating; Mindful awareness
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart rate variability biofeedback (Experimental): Heart rate variability biofeedback training will be administered via a smartphone app (Optimal HRV) that reads the participants' pulse rate through a Bluetooth connected photoplethysmography (PPG) sensor attached to the finger or thumb.
  Interventions: Behavioral: Heart rate variability biofeedback

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback — * 5 days of 3-min HRV readings to establish baseline HRV
  * After meeting with study personnel to review HRV biofeedback (BF) practice with the app, participants will be asked to begin HRV BF training for 5 min a day
  * Participants will increase the length of HRV BF training by 5 min every few days until they reach 20 min a day of HRV BF training
  * Participants will aim for 20 min of daily HRV BF training for 6 consecutive wks out of the 8-wk total BF training protocol
  * Study personnel will follow the participants' progress with training via the online portal provided through the Optimal HRV app and have brief (15-min) check-in appts. with participants to discuss how they are experiencing HRV BF, what they find helpful, and barriers to their practice if they are having difficulties
  * After completing the 8-wks of BF training (including 2 wks of 5-min titrations to the full 20-min protocol), participants will be asked to take 3-min HRV readings for 5 days to assess post-intervention HRV

SUMMARY:
As a result of the COVID-19 pandemic, the degree of burnout and consequential negative psychological effects experienced by healthcare providers has been substantially exacerbated. Heart rate variability (HRV) biofeedback has long been used to assist with a wide variety of stress-related concerns. Building on evidence that HRV biofeedback has the potential to improve wellbeing, the purpose of this study is to pilot test and determine the feasibility of implementing a digital HRV biofeedback tool to improve disordered eating, mindful self-care (i.e., self-compassion, body appreciation, etc.), and perceived stress in healthcare providers. In addition to assessing acceptability and feasibility of the HRV biofeedback tool, the investigators will aim to establish 'proof-of-concept' for a conceptual model consisting of potential psychological constructs underlying the mechanisms of change for the intervention-namely mind-body awareness (i.e., interoception) and resilience. Our primary recruitment pool will include healthcare providers who reported elevated eating distress as a participant in an ongoing observational study of the health effects of theCOVID-19 pandemic on essential workers (CHAMPS).

DETAILED DESCRIPTION:
Previous research suggests healthcare professionals may be a population at high-risk for disordered eating. As a result of the COVID-19 pandemic, the degree of burnout and consequential negative psychological effects experienced by healthcare providers has been substantially exacerbated. In fact, in an ongoing study of essential workers during the COVID-19 pandemic, the investigators found over a third of nursing professionals endorsed clinically significant disordered eating. With the clear evidence showing a psychological toll of the COVID-19 pandemic among healthcare workers globally, addressing their wellbeing with feasible at-home interventions is a priority.

Heart rate variability (HRV) biofeedback has long been used to assist with a wide variety of stress-related concerns, including depression and anxiety (Lehrer et al., 2020), both conditions that commonly co-occur with disordered eating. Research suggests interoception (i.e., the capacity to detect and respond to signals from the body), is disrupted in those with eating disorders (Martin et al., 2019). While there is relatively sparse evidence on the relationship between HRV and interoception (Pinna & Edwards, 2020), it is theoretically plausible that superior interoception would predict improved vagal tone (i.e., parasympathetic activity) as measured by HRV. Moreover, data on HRV and disordered eating is mixed, and poorly understood (Watford et al., 2020). The present research seeks to begin addressing this gap in knowledge through a pilot feasibility study designed to initiate proof-of-concept for the development of a conceptual model.

Specifically, the study aims to:

1. assess the feasibility of implementing a digitally based HRV biofeedback protocol
2. assess the acceptability and usability of HRV biofeedback in healthcare providers with elevated disordered eating
3. examine signals of efficacy to begin building a conceptual model of the potential mechanisms underlying change in outcomes
4. test whether there is a relationship between intervention engagement/adherence and change in outcomes.

Participants will be recruited from a registry of healthcare providers enrolled in an ongoing study of the health effects of working during the COVID-19 pandemic (unless recruitment goals are not met using this method). This single arm feasibility pilot will provide the data to help determine the acceptability of using a smartphone based HRV biofeedback training tool as an intervention for this population and guide the refinement of the conceptual model being developed. By establishing feasibility and proof-of-concept, the study will build upon a limited body of work and establish an important first step towards understanding intervention dosing and signals of efficacy for aiding with disordered eating and related mind-body factors in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Ability to speak and read English
3. Previously enrolled in the protocol titled "COVID-19 CHAMPS study" (IRB-FY2020-215) (ClinicalTrials.gov: NCT04370821)
4. Willing to be contacted about other studies (i.e., CHAMPS study participants who agreed to be contacted about future research opportunities)
5. Works in the healthcare professions
6. Elevated eating distress as indicated by Loss of Control Eating scores above the median of 2 in this cohort.
7. Owns either an iPhone or Android smartphone for running the app involved in the intervention

Exclusion Criteria:

1. History of a heart transplant or a pacemaker.
2. Uncontrolled kidney disease
3. Uncontrolled diabetes
4. Heart failure
5. COPD (Chronic Obstructive Pulmonary Disease)
6. Use of tricyclic antidepressant (e.g., nortriptyline, amitriptyline) above 75 mgs daily
7. Use of illicit stimulants (e.g., cocaine) or narcotic drugs
8. Inability to perform study protocol (self selected)
9. Current use of HRV biofeedback training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Pre-enrollment: | Consent interview/Baseline assessment - Week 0
  Measured by calculating the proportion of the people contacted who initially agree to participate in the study, defined as individuals who complete the baseline assessment following consent.
  This will assess feasibility to establish interest in HRV biofeedback among eligible participants from the CHAMPS registry.
Full enrollment: | Participant receipt of study device and initial study visit - Week 2
  Measured by calculating the proportion of the people who pre-enroll in the study who complete their first study visit that introduces the use of the HRV biofeedback app.
  This will assess feasibility to fully enroll participants in the HRV biofeedback protocol once they have agreed to participate and receive the device.
Engagement/adherence to protocol | Begins as soon the participant begins biofeedback training through the end of HRV biofeedback intervention - 8 weeks total
  Measured by calculating: a) the proportion of the fully enrolled participants meeting pre-determined study engagement criteria (i.e., =>28 days of the 42 where a minimum of 10 minutes of biofeedback is completed), and b) the total number of minutes of biofeedback training logged over the 8-week protocol.
  This will assess intervention's acceptability and serve as a measure of participant engagement
  *There is a change in this section from what was originally posted. The PI noticed a discrepancy between Aims stated on the funded grant proposal and ClinicalTrials.gov record therefore we fixed ClinicalTrials.gov so that it reflected the grant's Aims statement.
Attrition/Drop out | Training visit through final check-in and post-intervention assessments (approximately 10 weeks of study involvement
  Measured by calculating the proportion of fully enrolled participants who complete the pilot study.
  This is to assess feasibility of program implementation.
Usability | post-intervention assessment (approximately 8 weeks after HRV biofeedback training visit)
  Measured by calculating: a) the proportion of participants who rate HRV biofeedback practice as at least "moderately useful" (=>3 on a 1-5 Likert scale), and b) the proportion of participants who are at least "likely" (=>4 on a 1-5 Likert scale) to continue with their HRV biofeedback once the study ends.
  This is to assess the usability of HRV biofeedback in this population.

SECONDARY OUTCOMES:
Variation in disordered eating attitudes and behaviors | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit
  Measured using the Eating Disorder Examination-Questionnaire 7-itemBrief, (EDE-Q7 Range: 0-6, higher scores indicate worse outcome)
Variation in disordered eating attitudes and behaviors | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit
  Measured using the Loss of Control Eating Scale-7 item Brief (LOCES-Brief Range: 1-5, higher scores indicate worse outcome)
Variation in perceived stress | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Perceived Stress Scale, (PSS Range: 0-40, higher scores indicate worse outcome)
Variation in mindful self-care | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Mindful Self-Care Scale, (MSCS Range: depends on dimension, higher scores indicate better outcome)
Variation in interoception | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Multidimensional Assessment of Interoceptive Awareness - Version 2, (MAIA-v2 Range: 0-5, higher scores indicate better outcome)
Variation in interoception | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Hunger and Satiety subscale of the Intuitive Eating Scale-2 (IES-2 Range: 1-5, higher scores indicate better outcome)
Variation in body appreciation | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Body Appreciation Scale-2 (BAS-2 Range: 1-5, higher scores indicate better outcome)
Variation in resilience | baseline, midpoint (1 month after HRV biofeedback training visit), post intervention (2 months after HRV biofeedback training visit)
  Measured using the Sense of Coherence Scale Revised (SOC-R Range: depends on dimension, higher scores indicate better outcome)
Variation in HRV | baseline, post intervention (approximately 10 weeks after baseline assessment)
  Measured using the average daily RMSSD pre and post HRV biofeedback training

CONTACTS AND LOCATIONS:
Overall Officials: Janell Mensinger, PhD, Principal Investigator — Villanova University
Locations (1):
- Villanova University, Villanova, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators who contact the PI after establishing terms of use and collaborative agreement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When available

REFERENCES:
- [Background] Lehrer P, Kaur K, Sharma A, Shah K, Huseby R, Bhavsar J, Sgobba P, Zhang Y. Heart Rate Variability Biofeedback Improves Emotional and Physical Health and Performance: A Systematic Review and Meta Analysis. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):109-129. doi: 10.1007/s10484-020-09466-z. PMID 32385728
- [Background] Martin E, Dourish CT, Rotshtein P, Spetter MS, Higgs S. Interoception and disordered eating: A systematic review. Neurosci Biobehav Rev. 2019 Dec;107:166-191. doi: 10.1016/j.neubiorev.2019.08.020. Epub 2019 Aug 24. PMID 31454626
- [Background] Pinna T, Edwards DJ. A Systematic Review of Associations Between Interoception, Vagal Tone, and Emotional Regulation: Potential Applications for Mental Health, Wellbeing, Psychological Flexibility, and Chronic Conditions. Front Psychol. 2020 Aug 5;11:1792. doi: 10.3389/fpsyg.2020.01792. eCollection 2020. PMID 32849058
- [Background] Watford TS, Braden A, O'Brien WH. Resting state heart rate variability in clinical and subthreshold disordered eating: A meta-analysis. Int J Eat Disord. 2020 Jul;53(7):1021-1033. doi: 10.1002/eat.23287. Epub 2020 May 21. PMID 32437089
- [Derived] Mensinger JL, Weissinger GM, Cantrell MA, Baskin R, George C. A Pilot Feasibility Evaluation of a Heart Rate Variability Biofeedback App to Improve Self-Care in COVID-19 Healthcare Workers. Appl Psychophysiol Biofeedback. 2024 Jun;49(2):241-259. doi: 10.1007/s10484-024-09621-w. PMID 38502516